CLINICAL TRIAL: NCT05529329
Title: Clinical Outcome of Zirconia Versus Lithium Di-silicate Overlays Restorations for Restoring Vital Young Permanent First Molar Teeth Affected With Moderate Form of Molar Incisor Hypomineralization: Randomized Clinical Trial
Brief Title: Zirconia Versus Lithium Di-silicate Overlays for Restoring Hypomineralized Molars Affected With MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, AMMohammed, lecturer of Pediatric dentistry, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-PD-21-08
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Molar Incisor Hypomineralization
Keywords: MIH - zironia - Lithium Disilicate - Overlays
MeSH Terms: conditions — Molar Hypomineralization | interventions — Denture, Overlay

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (Z) (Active Comparator): patients received zirconia restorations group
  Interventions: Procedure: overlay
- Group (EC) (Experimental): patients received IPS E.max Cad restorations group
  Interventions: Procedure: overlay

INTERVENTIONS:
Procedure: overlay — Lithium Disilicate partial coverage of hypo-mineralized defected enamel
  Other Names: Zirconia partial coverage of hypo-mineralized defected enamel

SUMMARY:
the study evaluate the clinical outcome of zirconia versus lithium disilicate overlays restorations for restoring vital young permanent first molar teeth affected with moderate form of molar Incisor hypomineralization: randomized clinical trial.

DETAILED DESCRIPTION:
To compare the one-year clinical outcome of zirconia versus lithium disilicate overlays restorations. Materials and methods: Twenty patients were distributed into two groups in relation to the material used for the fabrication of overlays restorations; group (Z) (n=10): patients received zirconia restorations, group (EC): patients received IPS E.max Cad restorations. Clinical and radiographic evaluations of these restorations were carried out at base line (1 week), 3, 6 and 12 months after cementation using FDI World Dental Federation criteria

ELIGIBILITY:
Inclusion Criteria:

* Children's age ranging from 10 to 15 years old.
* Existence of large carious lesion in young permanent first molar teeth associated with weak cusps.
* Signs of vital pulp without symptoms of pulpitis.
* Presence of antagonists and adjacent teeth and occlusal contacts with good level of oral hygiene.
* Children should be able to physically and psychologically tolerate conventional restorative procedures.

Exclusion Criteria:

* Children with poor oral hygiene and symptoms of pulpitis.
* Children suffer from parafunctional habits.
* Children with any debilitating systemic disorder.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome | one year
  compare the one-year clinical outcome of zirconia versus lithium disilicate overlays
  restoration of vital young permanent first molar teeth affected with moderate form of Molar Incisor Hypomineralization
Restoration Evaluation | one year
  Restorations were assessed clinically using dental explorer, mirror and radiographically according to FDI World Dental Federation criteria over one-year period at (base line "1 week", 3, 6 and 12 months) afterward cementation. There were three assessment categories (esthetics, function, biological) each with five subcategories. From best to worst, the subcategories were: (1) clinically excellent, (2) clinically good, (3) clinically sufficient, (4) clinically not sufficient but repairable and (5) clinically unacceptable. Assessment with category (5) was rated as a clinical failure. Statistical analysis for baseline and follow-up criteria was performed with Wilcoxon-Test (p<0.05) (SPSS; IBM,Chicago, IL).

CONTACTS AND LOCATIONS:
Overall Officials: alaa F mohammed, Ph. D, Principal Investigator — Al-Azhar University- faculty of dentistry
Locations (1):
- Al-Azhar University, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Twenty patients were distributed into two groups in relation to the material used for the fabrication of overlays restorations; group (Z) (n=10): patients received zirconia restorations, group (EC): patients received IPS E.max Cad restorations. Clinical and radiographic evaluations of these restorations were carried out at base line (1 week), 3, 6 and 12 months after cementation using FDI World Dental Federation criteria
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: one year
Access Criteria: alaaaldehna.26@azhar.edu.eg